CLINICAL TRIAL: NCT05480163
Title: Acoustic and Volumetric Measurements in Order to Objectify Bronchial Congestion in Patients With Obstructive Respiratory Pathologies Within the Framework of Their Management in Respiratory Physiotherapy for Decongestion
Acronym: MUKROBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association des Réseaux Bronchiolite (Unknown)
Collaborators: Laboratoire Système et Matériaux pour la Mécatronique (SYMME) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUKROBS; 2021-A02143-38 (Other: ID-RCB)
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measurement records in COPD patients (Experimental): 1. The subject is informed of the procedure, his or her rights, and the use of the data collected (including the video recording of the session)
  2. Pre-session clinical assessment by the physiotherapist
  3. Installation of the Sybille waistcoat on the patient
  4. First measurement phase: Recording of spirometry parameters, acoustics, movements (thoracic volumetry) for forced vital capacity (FVC) and LVC manoeuvres.
  5. Second phase of measurements:
     Treatment: the physiotherapist performs the session in the classical way. Recording of acoustic parameters, movements (thoracic volumetry).
  6. Third phase of measurements: Recording of spirometry, acoustics and movement parameters (thoracic volumetry) for FVC and LVC manoeuvres.
  7. Removal of measurement devices
  8. Post session evaluation by the physiotherapist.
  Interventions: Other: Measurement records
- Measurement records in control subject (Other): 1. The subject is informed of the procedure, his or her rights, and the use of the data collected (including the video recording of the session)
  2. Clinical assessment by the physiotherapist The subject answers the questionnaire
  3. Installation of the Sybille waistcoat on the patient
  4. Measurement phase: Recording of spirometry, acoustics, movements (thoracic volumetry) for FVC and LVC manoeuvres.
  5. Removal of measurement devices
  Interventions: Other: Measurement records

INTERVENTIONS:
Other: Measurement records — Recordings of spirometry, acoustics, movement (chest volumetry) parameters for FVC and LVC exercises.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic respiratory disease defined by permanent airway obstruction. In this disease, a large part of the muscular work is taken up by breathing (fight against bronchial, parietal or fibrous resistances of the pulmonary tissue, reduction of the exchange surface), requiring a physiotherapeutic care.

Physiotherapy management of "respiratory rehabilitation" includes 4 items: respiratory therapy for decongestion, muscle strengthening, improvement of endurance and therapeutic education. In this context, the techniques of de-cluttering aim to decrease the hydrodynamic resistance of the bronchial tree. A systematic evaluation of the patient's condition is carried out by the practitioners to assess, at the time of the session, the bronchial congestion. In addition to their knowledge of the history of the patient they are following and the result of the oximetry measurement, practitioners use several indicators to assess the patient's bronchial congestion and define their therapeutic approach: cough, sputum, oximetry and peak expiratory flow, pulmonary auscultation. Sound expertise remains delicate: even the most educated human auditory system is not physiologically capable of detecting some of the relevant information. The current quantification criteria are therefore not very objective, depend on the practitioner's expertise and do not allow recommendations to be made on the conduct of the session during the follow-up of patients. Consequently, the objectification of bronchial congestion is clearly part of the process of improving management. In this context, the MUKROBS project seeks to objectify the bronchial congestion of COPD patients during their management by means of respiratory physiotherapy techniques of de-congestion by means of expiratory flow modulation techniques.

The Sybille device, designed, developed and validated in the framework of a previous project funded by the ANR VirtualChest, allows continuous, non-invasive and simultaneous measurements of sound and displacement information at specific points of the thoracic cage.

DETAILED DESCRIPTION:
COPD is a chronic respiratory disease defined by permanent airway obstruction. Epidemiological data are scarce: the prevalence is difficult to estimate because of underdiagnosis and the difficultý to perform respiratory function tests (RFTs) in epidemiological studies. It is estimated at 7.5% in a population over 45 years of age, with the incidence appearing to stabilize in men and increase in women. Furthermore, in 2018, 25.4% of adult patients had daily tobacco use. In 2014, 81,600 individuals were on long-term disability (LTD) for chronic bronchitis without specifics. The 2017 report by the Directorate for Research, Studies, Evaluation and Statistics (DREES) on the health status of the population in France shows that: in 2013, approximately 19,000 deaths were related to COPD, 48% of which were due to the initial cause; the crude mortality rateś related to COPD were 96/100,000 adults aged 45 years or older in men and 41/100,000 in women ; in 2014, the annual number of hospitalizations for COPD exacerbation ranged from 100 000 to 160 000, depending on the indicator; crude hospitalization rates were 31/10 000 in men and 15.4/10 000 in women, with the highest rates (>20%) in the northern and eastern regions of France and in Reunion. Standardized hospitalization rates have increased́ since 2000, by 2% per year in men and 5% per year in women. The average direct costs of COPD increase with the level of severitý of the disease and rise on average from €7,628 per year for the least severe patients to €20,747 per year for patients on oxygen therapy.

In this condition, a large part of the muscular work is taken up by breathing (fight against bronchial, parietal or fibrous resistances of the lung tissue, decrease of the exchange surface), requiring physiotherapeutic management.

The physiotherapeutic treatment "respiratory rehabilitation", includes 4 items: respiratory physiotherapy for decongestion, muscular strengthening, improvement of endurance and therapeutic education. Within this framework, the techniques of de-cluttering are intended to decrease the hydrodynamic resistance of the bronchial tree. A systematic evaluation of the patient's condition is carried out by the practitioners to assess, at the time of the session, the bronchial congestion. In addition to their knowledge of the history of the patient they are following and the result of the oximetry measurement, practitioners rely on several indicators to assess the patient's bronchial congestion and define their therapeutic approach: cough, sputum, oximetry and peak expiratory flow, pulmonary auscultation which provides sound information, and a call maneuver which allows a subjective assessment of the volumes that can be mobilized thanks to haptic information.

Sound expertise remains delicate: even the most educated human auditory system is not physiologically capable of detecting some of the relevant information. Multiple pathological breath sounds are referenced in the literature, for which different classifications exist, based on their frequency characteristics, their sound waveforms and their durations.

As for the haptic evaluation of thoracic compliance, it also requires a strong experience of the practitioner.

The current quantification criteria are therefore not very objective, depend on the practitioner's expertise and do not allow recommendations on the conduct of the session during the follow-up of the patients. Therefore, the objectification of bronchial congestion is clearly part of the improvement of the management of KR (Assess, Anticipate, Prevent, Treat). The design of specific tools dedicated to the quantified monitoring of relevant parameters of the lung condition is of definite interest to achieve these objectives.

In this context, the MUKROBS project seeks to objectivize the bronchial congestion of COPD patients, during their management by respiratory physiotherapy techniques of de-congestion by means of modulation of the expiratory flow.

The Sybille device, designed, developed and validated in the framework of a previous project funded by the ANR VirtualChest, allows continuous, non-invasive and simultaneous measurements of sound and displacement information at specific points of the thoracic cage. The investigators will conduct a measurement campaign in the context of follow-up in private practice. The measurements will be analyzed with numerical methods specifically developed in order to achieve an automatic identification of pathological respiratory sounds. The investigators will also try to localize bronchial obstructions and to correlate them with respiratory volume variations measured before, during and after the management session.

ELIGIBILITY:
Inclusion Criteria:

Control group

* Patient with no known respiratory pathology and a normal forced expiratory volume at one second (FEV1) /FVC ratio normal for age and sex (chart).

COPD group

* Patients diagnosed with COPD, post exacerbations and/or post hospitalisation with chronic congestion

Exclusion Criteria:

Control group

* Smoker or former smoker (less than 6 years of cessation)
* Prolonged or repeated exposure to gases, dusts, fumes, vapours in the context of professional activities
* Respiratory pathology
* Pacemaker or heart battery wearers
* Cognitive disorders that do not allow for informed consent
* Prostheses or metallic materials (vascular clip, neuro-stimulator, insulin pump, various implants, etc.)
* Chest pain context
* Spinal orthopaedic disorders not compatible with the device (cypho scoliosis etc...)
* Opposition of the patient
* BMI >30
* History of hospitalization for coronavirus

COPD group :

* Refusal to transfer image rights
* Haemoptysis
* Pacemaker or heart battery wearers
* Cognitive impairment that does not allow for informed consent
* Prostheses or metallic devices (vascular clip, neuro-stimulator, insulin pump, various implants)
* Presence of oppressive chest pain
* Neurological pathologies (Parkinson's, etc.)
* Paradoxical breathing
* Spinal orthopaedic disorders not compatible with the device (cypho scoliosis etc...)
* Opposition of the patient
* BMI >30
* History of hospitalization for coronavirus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Scoring of respiratory congestion | 75 minutes
  Comparison of the scoring of respiratory congestion status assessed by expert physiotherapists and by the Sybille device.

SECONDARY OUTCOMES:
Respiratory volumes in COPD group | 75 minutes
  Respiratory volumes, before and after decongestion manoeuvres, obtained by spirometer in the COPD group.
Volumes calculated from the displacements | 75 minutes
  The volumes calculated from the displacements recorded by the Sybille device of 8 points located on the rib cage, before, during and after the decongestion manoeuvres, in the COPD group.
Respiratory volumes in control group | 40 minutes
  Respiratory volumes obtained by the spirometer in the control group.
Volumes calculated in control group | 40 minutes
  The volumes calculated from the displacements recorded by the Sybille device of 8 points located on the rib cage, in the control group.
Rates by type of breath sounds | 75 minutes
  The rates by type of breath sounds before, during and after the de-cluttering manoeuvres from the sounds recorded by the Sybille device, in the COPD group.
Haptic sensations and the number and type of pathological breath | 75 minutes
  The haptic sensations and the number and type of pathological breath sounds recorded during auscultations by the expert physiotherapists, and which are recorded in a questionnaire, for the COPD group
Practitioners' treatment strategies | 75 minutes
  Practitioners' treatment strategies described by Flanagan's critical incident method, in the COPD group.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Physiotherapy practice of Mr TORRES, Annecy
  - Physiotherapy practice of Mr. Jean-Charles LAPORTE, Paris